CLINICAL TRIAL: NCT03375684
Title: Effects of Inspiratory Muscle Training on Postural Stability, Balance, Pulmonary Function and Functional Capacity in Children With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Melih Zeren, Lecturer, MSc, PT, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bvumzeren01
Record Dates: First submitted 2017-12-06; First posted 2017-12-18 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Inspiratory Muscle Training; Chest Physiotherapy; Balance; Postural Stability; Pulmonary Function Test; 6-Minute Walk Test
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients in this group will receive conventional chest physiotherapy, two times a day, 7 days a week for 8 weeks. One exercise session will be supervised in a clinic per week, other sessions will be performed at home.
  Interventions: Other: Conventional chest physiotherapy
- Training Group (Experimental): In addition to conventional chest physiotherapy programme, patients in this group will also receive inspiratory muscle training for 15 minutes, twice a day, 7 days a week for 8 weeks. One exercise session will be supervised in a clinic per week, other sessions will be performed at home.
  Interventions: Other: Conventional chest physiotherapy; Other: Inspiratory muscle training

INTERVENTIONS:
Other: Conventional chest physiotherapy — Programme will include diaphragmatic breathing exercise, thoracic expansion exercises, incentive spirometer exercise (Triflo), oscillatory PEP (Flutter), postural drainage and coughing tecniques.
Other: Inspiratory muscle training — Threshold IMT device will be used for the training. Training intensity will set at 30% of the maximum inspiratory pressure.
  Arms: Training Group

SUMMARY:
It is extensively reported in the literature that patients with chronic obstructive lung disease may have impairments in balance and postural control which further increase the disease burden. Mechanisms related to these impairments include, but are not limited to increased work of breathing, diaphragm weakness, peripheral muscle weakness and systemic inflammation. Since the similar symptoms are reported for the children with cystic fibrosis, it is hypothesized that balance and postural control may also be compromised in these patients. Inspiratory muscle training (IMT) is shown to improve diaphragm strength and pulmonary function. Considering the relation between diaphragm which is one of the core muscles, and balance, IMT may also have an impact on postural control and balance alongside the standard clinical parameters such as respiratory muscle strength, pulmonary function and functional capacity in these patients. Thus, the aim of this study was to investigate the effects of inspiratory muscle training and conventional chest physiotherapy on postural stability, balance, pulmonary function and functional capacity in children with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis diagnosis
* Stable clinical condition (no exacerbation in last 4 weeks)

Exclusion Criteria:

* Documented diagnosis of vestibular, neurological or orthopedic disorders which may affect balance and mobility
* Subjects previously involved in exercise training or physiotherapy programs

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline postural stability test score in Biodex Balance System SD at 8 weeks | Eight weeks
Change from baseline limits of stability test score in Biodex Balance System SD at 8 weeks | Eight weeks
Change from baseline sensory integriation and balance test score in Biodex Balance System SD at 8 weeks | Eight weeks
Change from baseline Forced Vital Capacity (FVC) at 8 weeks | Eight weeks
Change from baseline Forced Expiratory Volume in 1 second (FEV1) at 8 weeks | Eight weeks
Change from baseline Peak Expiratory Flow (PEF) at 8 weeks | Eight weeks
Change from baseline maximum inspiratory pressure at 8 weeks | Eight weeks
Change from baseline maximum expiratory pressure at 8 weeks | Eight weeks
Change from baseline distance covered in six-minute walk test at 8 weeks | Eight weeks

SECONDARY OUTCOMES:
Change from baseline m. quadriceps strength at 8 weeks | Eight weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif Universitesi, Department of Physiotherapy and Rehabilitation, Istanbul, Eyup, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zeren M, Cakir E, Gurses HN. Effects of inspiratory muscle training on postural stability, pulmonary function and functional capacity in children with cystic fibrosis: A randomised controlled trial. Respir Med. 2019 Mar;148:24-30. doi: 10.1016/j.rmed.2019.01.013. Epub 2019 Jan 28. PMID 30827470